CLINICAL TRIAL: NCT05663372
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Efez 50 mg Eplerenone Film-coated Tablets Versus INSPRA® 50 mg Eplerenone Film-coated Tablets, in Healthy Adult Male and Female Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Test and Reference 50 mg Eplerenone Film-coated Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Darnitsa Pharmaceutical Company (Industry)
Collaborators: ACDIMA Biocenter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EPL01-E
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Bioequivalence; Healthy Subjects
Keywords: bioequivalence; eplerenone; healthy subjects; pharmacokinetics
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Intervention Model Description: Two-period, two-sequence, two-way, crossover, single dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efez (Test) (Experimental): A single oral dose of the test product Efez 50 mg eplerenone film-coated tablets.
  Interventions: Drug: Efez 50 mg eplerenone film-coated tablets
- INSPRA® (Active Comparator): A single oral dose of the reference product INSPRA® 50 mg eplerenone film-coated tablets.
  Interventions: Drug: INSPRA® 50 mg eplerenone film-coated tablets

INTERVENTIONS:
Drug: Efez 50 mg eplerenone film-coated tablets — Oral, mineralocorticoid receptor antagonist, a blocker of aldosterone
  Arms: Efez (Test)
Drug: INSPRA® 50 mg eplerenone film-coated tablets — Oral, mineralocorticoid receptor antagonist, a blocker of aldosterone
  Arms: INSPRA®

SUMMARY:
This study is a comparative bioavailability study performed to assess bioequivalence between Test medicinal product (Efez 50 mg eplerenone film-coated tablets manufactured by PrJSC "Pharmaceutical firm "Darnitsa", Ukraine) and Reference medicinal product (marketed medicinal product INSPRA® 50 mg eplerenone film-coated tablets, Marketing Authorisation Holder: Pfizer Europe MA EEIG, Belgium) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is Caucasian & aged between eighteen to fifty years (18 - 50), both inclusive.
2. The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
3. The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
4. The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator.
5. The subject tested negative for hepatitis B (HBsAg), hepatitis C (HCVAb), human immunodeficiency virus (HIVAb) & COVID-19 (PCR) test.
6. There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
7. The subject is able to understand and willing to sign the informed consent form.
8. For female subjects: a negative pregnancy test must be confirmed, and if sexually active, at least 4 weeks of highly effective contraceptive method must be used prior to IMP administration and throughout the study progress until last visit; highly effective methods comprise hormonal contraceptives, intrauterine devices IUDs, sexual abstinence or vasectomized partner (success of vasectomy was medically proven). For subjects using a hormonal contraceptive method, a barrier form of contraception should be combined with the hormonal contraception.
9. The subject has normal cardiovascular system & ECG recording.
10. The subject kidney and liver (AST & ALT enzymes) functions tests are within normal range.
11. The subject blood pressure is ≥ 110/70 mmHg before dosing.
12. The subject has normal serum creatinine and potassium levels on screening (before 24 hours of admission).
13. The subject HbA1c test result is within normal range.

Exclusion Criteria:

1. Subject is a smoker or an ex-smoker with a non-smoking history of less than 6 months.
2. The subject has suffered an acute illness one week before dosing.
3. The subject has a history of or concurrent abuse of alcohol.
4. The subject has a history of or concurrent abuse of illicit drugs.
5. The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
6. The subject has been hospitalized within three months before the study or during the study.
7. The subject is on special diet (for example subject is vegetarian).
8. The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 36 hours after dosing in all study periods.
9. The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
10. The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
11. The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
12. The subject has donated blood within 80 days before first dosing.
13. The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
14. The subject has consumed drugs or foodstuffs that may affect pharmacological or pharmacokinetic properties of eplerenone (for example: strong CYP3A inhibitors (e.g., ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, and nelfinavir), potassium supplements or potassium-sparing diuretics (e.g., amiloride, spironolactone, or triamterene), ACE inhibitors and angiotensin II receptor antagonists, lithium or NSAIDs) two weeks before dosing, during the study and two weeks after dosing.
15. Pregnant; with positive serum pregnancy test or breast-feeding female subjects.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Blood sampling for pharmacokinetic analysis covered up to 36 hours post-dose.
  The Cmax value is based on the eplerenone plasma concentration.
Area under the concentration-time curve from time zero to the last quantifiable concentration (t) | Blood sampling for pharmacokinetic analysis covered up to 36 hours post-dose.
  The AUC0-t is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (t) and is based on the eplerenone plasma concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- ACDIMA Center for Bioequivalence and Pharmaceutical Studies, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No